CLINICAL TRIAL: NCT01129089
Title: Acceptability of Lipid-based Nutrient Supplements (LNS) and Micronutrient Powder (MNP) for Women and Infants in Bangladesh
Brief Title: Acceptability of Nutrient Supplements Among Women and Children in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 273918; 4001-UCD-00 (Other Grant/Funding Number: Food and Nutrition Technical Assistance II (FANTA-2))
Record Dates: First submitted 2010-05-13; First posted 2010-05-24 (Estimated); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Malnutrition
Keywords: Acceptability; Lipid-based nutrient supplements; Micronutrient powder; Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LNS-PLW (Experimental): There will be 48 pregnant or lactating women (PLW) in this arm. They will be randomized to receive cumin flavored LNS-PLW or LNS-PLW with no added flavor on day 2. On day 3, the PLW getting a test-dose of cumin flavored LNS-PLW on day 2 will receive LNS-PLW with no added flavor and the PLW getting a test-dose of LNS-PLW with no added flavor on day 2 will receive cumin flavored LNS-PLW.
  Interventions: Dietary Supplement: Lipid-based nutrient supplement
- LNS-Child (Experimental): There will be 48 infant and young children(IYC) in this arm. They will be randomized to receive cardamom flavored LNS-Child or LNS-Child with no added flavor on day 2. On day 3, the IYC getting a test-dose of LNS-Child with no added flavor on day 2 will receive cardamom flavored LNS-Child and the IYC getting a test-dose of cardamom flavored LNS-Child on day 2 will receive LNS-Child with no added flavor.
  Interventions: Dietary Supplement: Lipid-based nutrient supplement
- MNP-Child (Experimental): There will be 48 infant and young children(IYC) in this arm. They will receive MNP on day 2 and day 3.
  Interventions: Dietary Supplement: Micronutrient powder

INTERVENTIONS:
Dietary Supplement: Lipid-based nutrient supplement — Lipid-based nutrient supplement for pregnant and lactating women
  Other Names: LNS
  Arms: LNS-PLW
Dietary Supplement: Lipid-based nutrient supplement — Lipid-based nutrient supplement for infant and young children
  Other Names: LNS
  Arms: LNS-Child
Dietary Supplement: Micronutrient powder — Micronutrient powder for infant and young children
  Other Names: MNP; Sprinkles
  Arms: MNP-Child

SUMMARY:
The study aims to confirm the acceptability of lipid-based nutrient supplements (LNS) for use as nutritional supplements for pregnant and lactating women (PLW) or infants and young children (IYC) and micronutrient powder (MNP) for use as nutritional supplements for infants and young children in Bangladesh.We hypothesized that at least 75 percent of the test dose of LNS and MNP offered to PLW and IYC will be consumed by them.

DETAILED DESCRIPTION:
The study will be conducted in three steps. Step 1 will be a test-feeding to compare the acceptability of each "version" of the LNS-child (LNS-child with cardamom flavor, LNS-child with no added flavor),LNS-PLW (LNS-PLW with cumin flavor, and LNS-PLW with no added flavor) and MNP to the others in terms of taste, smell and texture, as well as amount of the test-dose consumed. In Step 2, participants in the Phase 1 trial will receive a 2-week supply of one of the LNS products or MNP, which they will consume daily in their homes for 14 days under real-life conditions. In Step 3, focus group discussions will be held with participants to discuss different aspects of infant and child feeding and discuss best ways for the LNS or MNP product to be used in the context of Bangladesh.

ELIGIBILITY:
Inclusion criteria for LNS-PLW arm:

* Pregnant women in their second or third trimester (in case of third trimester pregnancy, the expected date of delivery is not within three weeks) or lactating women with a child between 3 days and 6 months of age
* At least 18 years of age
* No life-threatening pregnancy-related complications (e.g., pre-eclampsia, antepartum hemorrhage)
* Apparently healthy and not presently suffering from an acute illness (e.g., fever, diarrhea, acute respiratory tract infection)
* Living in the study area for at least 6 months
* Planning to remain in study area for at least the following three weeks.

Exclusion criteria for LNS-PLW arm:

* Known allergy to peanuts or other food products (as reported on the screening questionnaire)

Inclusion criteria for LNS-Child and MNP-Child arm:

* Children 6-24 months of age
* Consuming solid foods for at least the past 30 days
* Apparently healthy and not presently suffering from an acute illness (e.g., fever, diarrhea, acute respiratory tract infection)
* No known allergy to peanuts or other food products (as reported on the screening questionnaire by the mother/primary caregiver)[LNS-Child only]
* Planning to remain in study area for at least the following three weeks.

Exclusion criteria for LNS-Child and MNP-Child arm:

* Severely malnourished [mid-upper arm circumference (MUAC) < 115 mm]

Ages: 6 Months to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2009-12; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Proportion of test dose consumed | Day 2
  Mean consumption of the test dose of LNS for PLW, LNS for IYC and MNP for IYC on day 2 (First test dose)
Proportion of test dose consumed | Day 3
  Mean consumption of the test dose of LNS for PLW, LNS for IYC and MNP for IYC on day 3(Second test dose)

SECONDARY OUTCOMES:
Proportion of subjects liked the supplements | Day 2
  Using a five point Likert scale proportion of PLW and IYC liked the supplements will be acertained.
Proportion of subjects liked the supplement | Day 3
  Using a five point Likert scale proportion of PLW and IYC liked the supplements will be acertained.
Proportion of subjects liked the supplement | Day 8
  Using a five point Likert scale proportion of PLW and IYC liked the supplements will be acertained.
Proportion of subjects liked the supplement | Day 15
  Using a five point Likert scale proportion of PLW and IYC liked the supplements will be acertained.

CONTACTS AND LOCATIONS:
Overall Officials: Katnryn G Dewey, Ph.D., Principal Investigator — University of California, Davis; Malay K Mridha, MBBS,MPH, Study Director — University of Callifornia, Davis; Camila M Chaparro, Ph.D., Study Director — Academy for Educational Development
Locations (1):
- Fatejangpur, Chirirbandar, Dinajpur, Bangladesh